CLINICAL TRIAL: NCT02894359
Title: Computer Modelling of the Cervical Spine Movements in Cervical Dystonia
Acronym: STICOB
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SSA_2016_19
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Cervical Dystonia, Primary
Keywords: Cervical spine; Musculoskeletal imagery; computer modelling of cervical spine; ConeBeam.
MeSH Terms: conditions — Cervical Dystonia, Primary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- CD patients: 10 patients with a cervical dystonia
  Interventions: Device: cone beam imagery of cervical spine
- control subjects: 10 healthy patients
  Interventions: Device: cone beam imagery of cervical spine

INTERVENTIONS:
Device: cone beam imagery of cervical spine

SUMMARY:
Cervical dystonia (CD) is a syndrome characterized by sustained and/or phasic involuntary neck muscle activity causing abnormal head postures and movements. It is the most frequent form of adult focal dystonia. The distribution of dystonic muscles is unique for each patient, explaining the variety of patterns encountered.

The therapeutic management of CD is essentially local and symptomatic: Botulinum Neurotoxin injections and/or specific retraining therapy programmes. Therefore, analyzing the characteristics of abnormal head movements and identifying the dystonic muscles are the key points of these treatments.

To a better understanding of the posture and movement disorders of head and neck, we wish to establish a three-dimensional (3-D) computer model of cervical spine movements of ten healthy subjects built from images obtained with the "Cone Beam " system. Then we will compare the cervical posture and movements for each of ten CD patients matched in age and genre to the computer model. Comparison with patients' images in the axial plane reconstructed by computer with the 3-D computer model will lead to the description of various patterns of CD. Analysis of the musculoskeletal disturbances in CD should be a help to improve the localization of Botulinum Neurotoxin injection sites as well as retraining programmes.

ELIGIBILITY:
Inclusion Criteria:

* Tonic form of focal or segmental cervical dystonia (diagnostic confirmed by a neurologist specialized in movement disorders) for CD patients, or absence of CD for control subjects
* absence of treatment by botulinum neurotoxin, or last injection > 3 months
* age > 18 and < 71 years
* informed consent
* medical insurance coverage

Exclusion Criteria:

* CD mobile (clonic) and/or head tremor
* patient unable to sit without moving the head during the examination (x-ray pictures with cone beam)
* Other neurological disease with effect on the posture and/or movement of the cervical region
* Pain or traumatism of the cervical region requiring medical or surgical treatment in the preceding 6 months
* Pregnant or breast feeding patient
* Participation in another research with a potential impact on evaluation criteria
* patient under judiciary protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 CD patients without Botulinum neurotoxin injection in the preceding 3 months and 10 control subjects, age and gender matched.
  All subjetcts included in the study will undergo cervical spine imagery with the cone beam device (static and cervical rotation).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
comparison of bone marks positions (degrees) in patients ans control motions | baseline
  positions measured in degrees with computerized imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre BLETON, PhD, Study Chair — Fondation OPH A de Rothschild; Sophie SANGLA, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, France